CLINICAL TRIAL: NCT03702920
Title: Effects of Plasma Exchange With Human Serum Albumin 5% (PE-A 5%) on Short-term Survival in Subjects With "Acute-On-Chronic Liver Failure" (ACLF) at High Risk of Hospital Mortality
Brief Title: Short-term Survival of Subjects With Acute-on-chronic Liver Failure After Plasma Exchange With Human Serum Albumin 5%
Acronym: APACHE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to corporate business reasons only (non-safety related decision)
Sponsor: Grifols Therapeutics LLC (Industry)
Collaborators: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IG1407
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SMT+ PE-A 5% (Experimental): PE-A 5% will be performed using 5% albumin (Albutein 5%) as the main replacement fluid administered intravenously.
  Interventions: Biological: SMT + PE-A 5%
- Standard Medical Treatment (SMT) (Active Comparator): Standard medical treatment (SMT) will be administered according to institution standards.
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Biological: SMT + PE-A 5% — Plasma exchange treatment (PE-A 5%) will be performed using 5% albumin solution (Albutein 5%). Fresh frozen plasma will be given to prevent coagulopathy. IVIGs will be administered intravenously to prevent the development of hypogammaglobulinemia and infection.
  Other Names: Albutein 5%
  Arms: SMT+ PE-A 5%
Other: Standard Medical Treatment — Standard medical treatment according to the institution's standard practice
  Other Names: SMT
  Arms: Standard Medical Treatment (SMT)

SUMMARY:
This is a Phase 3, multicenter, randomized, controlled, parallel-group, open-label study to evaluate the effects of plasma exchange using human serum albumin 5% (PE-A 5%) in acute-on-chronic liver failure (ACLF) subjects. The study will involve approximately 40 study centers in the United States, Canada, and Europe with expertise in the management of subjects with ACLF.

Subjects with ACLF at a high risk of hospital mortality will be enrolled. The study will consist of a Screening Period during which subjects will be randomized (1:1) to receive either standard medical treatment (SMT) + PE-A 5% (treatment group) or SMT only (control group), followed by a Treatment Period, and a Follow-up Period.

The Treatment Period for subjects in the SMT+ PE-A 5% treatment group will be between 7 and 17 days, depending on ACLF evolution.

The Treatment Period for subjects in the SMT control group will be a minimum of 7 days for all subjects and up to 17 days depending on the ACLF evolution. Subjects in this group will receive SMT according to the institution's standards.

The Follow-up Period for subjects in both groups will be 90 days.

DETAILED DESCRIPTION:
Approximately 380 subjects with cirrhosis, ACLF, and high risk of hospital mortality (ACLF-1b, ACLF-2, or ACLF-3a) will be included in this study after obtaining written informed consent. In case of hepatic encephalopathy (HE), written informed consent will be obtained from a relative or a legally authorized representative if the subject is considered incompetent to consent.

Randomization of subjects will be stratified by region (European Union [EU] or North America [NA]) and the 3 ACLF grades (ACLF-1b, ACLF-2, or ACLF-3a). Within each stratum (ie, each unique combination of region and ACLF grade), subjects will be randomized in a 1:1 ratio into 2 treatment groups below:

* SMT+PE-A 5% (treatment group)
* SMT (control group)

SMT + PE-A 5% Treatment Group:

PE-A 5% will be performed using 5% albumin (Albutein® 5%) as the main replacement fluid administered intravenously. Fresh frozen plasma (FFP) will be given after each PE-A 5% session to prevent coagulopathy.

The exact number of sessions will be determined by the pattern of response (achieving complete response or no improvement/deterioration of ACLF) to PE-A 5% therapy. IVIGs will be administered to prevent the development of hypogammaglobulinemia and infection.

SMT Control Group:

The Treatment Period will be 7 days for all subjects and will be prolonged depending on subject's ACLF evolution to up to 17 days.

Subjects in both the SMT+ PE-A 5% treatment group and the SMT control group will be followed for 90 days after randomization. During the entire study, the safety of both groups will be monitored by a Data Safety Monitoring Board.

ELIGIBILITY:
Inclusion Criteria:

* Male or female cirrhotic subjects between 18 and 79 years of age.
* Subjects with ACLF-1b, ACLF-2, or ACLF-3a detected either at admission or during hospitalization (must be ACLF-1b, -2, or -3a within the Screening Period [a maximum of 10 days]).
* Willing and able to provide written informed consent or have an authorized representative able to provide written informed consent on behalf of the subject in accordance with local law and institutional policy.
* In case of HE, informed consent will be provided by a relative or a legally authorized representative if the subject is considered incompetent to consent.

Exclusion Criteria:

* Subjects without ACLF.
* Subjects with ACLF-1a or ACLF-3b (See Table 2-1 for ACLF grades) after the Screening Period.
* Subjects fulfilling inclusion criteria that improve to no ACLF or to ACLF-1a or worsen to ACLF-3b during the Screening Period (between initial evaluation and time of randomization).
* Subjects with ACLF for more than 10 days prior to randomization.
* Subjects with acute or subacute liver failure without underlying cirrhosis.
* Subjects with septic shock requiring use of norepinephrine (> 0.3 mcg/kg/min) or need for a second vasopressor (including terlipressin).
* Subjects with active bacterial or fungal infection: who have received less than 24h of appropriate antibiotic treatment.
* Subjects with severe respiratory failure with PaO2/FiO2 ≤200.
* Subjects with active or recent bleeding (unless controlled for >48 hours).
* Subjects with severe thrombocytopenia (≤20×109/L) (based on local laboratory assessment).
* Subjects with chronic renal failure and currently receiving hemodialysis.
* Evidence of current locally advanced or metastatic malignancy. Subjects with hepatocellular carcinoma within the Milan criteria (1 nodule ≤5 cm or 3 nodules ≤3 cm [Appendix 5]), non-melanocytic skin cancer, and controlled breast or prostate cancer, can be included).
* Subjects with severe chronic heart failure (New York Heart Association [NYHA] class III or IV).
* Subjects with severe pulmonary disease (Global Obstructive Lung Disease [GOLD] stage III or IV).
* Subjects with severe myopathy as defined clinically.
* Subjects with a known infection with human immunodeficiency virus (HIV) or have clinical signs and symptoms consistent with current HIV infection.
* Females who are pregnant, breastfeeding, or if of childbearing potential, unwilling to practice a highly effective method of contraception.
* Subjects with previous liver transplantation.
* Subjects receiving anti-platelet or anti-coagulant therapy (LMWH for DVT prophylaxis is allowed).
* Participation in another clinical study within at least 30 days prior to screening.
* Subjects with active drug addiction (exceptions: active alcoholism or marijuana).
* Subjects with a do-not-resuscitate order.
* In the opinion of the investigator, the subject may have compliance problems with the protocol and the procedures of the protocol.
* Subjects with current infection of COVID19, those who are less than 14 days post recovery or those who have clinical signs and symptoms consistent with COVID19 infection.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Time to death through Day 90 | Day 1 to Day 90
  Time to death through Day 90 after randomization of SMT+PE-A 5% versus SMT alone

SECONDARY OUTCOMES:
Time to transplant or death through Day 90 | Day 1 to Day 90
  Time to transplant or death through Day 90 after randomization of SMT+PE-A 5% versus SMT alone
Time to death through Day 28 | Day 1 to Day 28
  Time to death through Day 28 after randomization of SMT+PE-A 5% versus SMT alone

CONTACTS AND LOCATIONS:
Locations (40):
- United States (15):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Southern California Research Center, Coronado, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - University of Kansas, Kansas City, Kansas
  - Rutgers-New Jersey Medical School, Newark, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Mayo Clinic Rochester, Rochester, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - McGuire VA Medical Center, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Aurora Health Care, Inc., Milwaukee, Wisconsin
- Medical University of Vienna, Vienna, Austria
- Belgium (2):
  - Université libre de Bruxelles, Brussels
  - UZ Leuven - Campus Gasthuisberg, Leuven
- Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Hôpital Beaujon, Clichy
  - Centre Hépato-Biliaire - Hôpital Universitaire Paul Brousse, Villejuif
- Germany (5):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Frankfurt, Frankfurt
  - Hannover Medical School, Hanover
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Universitaet Muenchen, München
- Italy (5):
  - ASST Papa Giovanni XXIII, Bergamo
  - Milano Hospital Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Roma
- Portugal (2):
  - Centro Hospitalar Lisboa Norte, Lisbon
  - Centro Hospitalar do Porto, Porto
- Spain (4):
  - Hospital Universitario del Valle Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
- United Kingdom (3):
  - Royal Free NHS Foundation Trust Hospital, London
  - King's College Hospital NHS Foundation Trust, London
  - Nottingham University Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No